CLINICAL TRIAL: NCT04874376
Title: Clinical Study to Investigate Visual Performance, Contrast Sensitivity and Patient Satisfaction After Implantation of a Premium Monofocal Intraocular Lens
Brief Title: PMCF Retrospective Study Outcomes of a Premium Monofocal IOL
Acronym: PHY2110
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY2110
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular Lens; Premium; hydrophobic; IOL; monofocal
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOL retrospective data collection (Experimental): Experimental arm: Premium Monofocal intraocular lens.
  Interventions: Device: IOL implantation experimental (Isopure 1.2.3.)

INTERVENTIONS:
Device: IOL implantation experimental (Isopure 1.2.3.) — Implantation of Premium Monofocal Isopure 12.3 with retrospective data collection

SUMMARY:
Multicentric, retro- / prospective, open-label, observational PMCF study to investigate visual performance, contrast sensitivity and patient satisfaction after mono- or bilateral implantation of Isopure 1.2.3. intraocular lenses following cataract surgery.

The study treatment itself is not part of this observational clinical investigation. Only patients that already have been implanted with the device under investigation qualify for this retro- prospective observational clinical study.

DETAILED DESCRIPTION:
The study is a multicentric, retro- / prospective, open-label, observational PMCF study to investigate visual performance, contrast sensitivity and patient satisfaction after mono- or bilateral implantation of Isopure 1.2.3. intraocular lenses following cataract surgery.

The study treatment itself is not part of this observational clinical investigation. Only patients that already have been implanted with the device under investigation qualify for this retro- prospective observational clinical study.

Isopure 1.2.3. is CE approved and commercially available in the countries this clinical investgation is being carried out. The investigational device and all study products, including the devices used for the study examinations, will be used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the patient.

The study will be carried out in up to five clinical centers in Spain. The device under investigation (Isopure 1.2.3.) is a hydrophobic, glistening-free, acrylic Premium Monofocal intraocular lens (IOL) manufactured by the sponsor of this study, PhysIOL sa/nv.

Subjects participating in the trial will attend a total of maximum 1 study visit (from 120 days post-operative). This study visit will be minimum 20 days after the surgery of the 2nd eye. Subjects would have the option for unscheduled visits if required medically.

The primary performance endpoint is to show that the monocular Best Corrected Distance Visual Acuity (CDVA) measured in the study group is statistically non-inferior to outcomes of the monofocal parent lens Micropure 1.2.3. The comparative data is used from the latest Clinical Evaluation Report (CER) for the monofocal Micropure 1.2.3. lens. To avoid bias, only the first implanted eye will be considered for this calculation. Data interim analyses will be done after the last patient finished the 1 study visit postoperative examination to support the study publication plan.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female adults ages 45 years or older on the day of treatment that were mono- or bilaterally implanted with Isopure 1.2.3. intraocular lens minimum 120 days before the study visit;
* Maximum time between first and second eye treatment: 45 days (this accounts for bilateral implantations only);
* Capability to understand and sign an IRB approved informed consent form and privacy authorization;
* Clear intraocular media;
* Minimum set of retrospective preoperative and intraoperative data available as outlined in the examination matrix;
* Willing and able to conform to the study requirements.

Exclusion Criteria:

* • Age of patient <45 years at the day of surgery;
* Time between first and second eye treatment: >45 days (this accounts for bilateral implantations only);
* Subjects who underwent previous intraocular or corneal surgery other than IOL implantation;
* Subjects with diagnosed degenerative visual disorders (e.g. AMD or CME);
* Subjects in whom in-the-bag implantation was not possible;
* Subjects in whom surgical complications occurred (e.g. posterior rupture).
* Subjects showing glaucoma;

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
monocular Best Corrected Distance Visual Acuity (CDVA) under photopic light conditions on the first implanted eye. | From 120 days postoperative
  No statistically significant difference between the monocular CDVA from 4 months follow up visit when compared to the parent IOL (Micropure 1.2.3). A significance level of 0.025 or lower (p < 0.025) will be considered statistically significant. CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Bernabeu Arias, MD, Principal Investigator — HM Monteprincipe, HM Vallés, Madrid, Spain
Locations (6):
- Spain (6):
  - Oftalvist, Alicante, Alicante
  - Vithas, Alicante, Alicante
  - Clinica Baviera, Madrid
  - HM Monteprincipe, Madrid
  - HM Vallés, Madrid
  - Augenklinik, Palma de Mallorca, Multiple Locations

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605